CLINICAL TRIAL: NCT06950060
Title: AMPLIFI: Adaptive Modulation of Plasticity Through Lactate and Fitness Interventions
Acronym: AMPLIFI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Keith McGregor, Associate Professor, Director of Research, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-300014361
Record Dates: First submitted 2025-04-03; First posted 2025-04-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Stroke, Chronic; Aging; Cognitive Decline; Motor Dysfunction; Neuroplasticity
Keywords: Transcranial Magnetic Stimulation (TMS); Cortical Inhibition; Neuroplasticity; Aerobic Exercise; Motor Learning; Aging; Stroke Rehabilitation; Cortical Excitability; GABAergic Inhibition
MeSH Terms: conditions — Stroke; Bronchiolitis Obliterans Syndrome; Cognitive Dysfunction; Neurologic Manifestations | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Participants are randomized into one of four parallel groups: (1) aerobic exercise at lactate threshold, (2) moderate intensity exercise, (3) low-intensity aerobic exercise, or (4) education-only control. Outcomes are assessed at multiple time points to examine changes in cortical inhibition, motor performance, and cognitive function.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aerobic Exercise at Lactate Threshold (Experimental): Participants complete a 20-minute aerobic cycling session at individually prescribed intensity to achieve lactate threshold, based on VO2 max and blood lactate data. This condition is designed to induce metabolic stress and engage neuromodulatory pathways related to cortical plasticity. Participants complete TMS and motor learning tasks before and after the intervention.
  Interventions: Behavioral: High intensity cycling
- Low-Intensity Aerobic Exercise (Active Comparator): Participants complete a 20-minute cycling session at a light workload, below lactate threshold. This condition controls for movement and engagement without significant metabolic challenge. TMS and motor learning outcomes are assessed pre- and post-intervention.
  Interventions: Behavioral: Low-intensity cycling
- Education Control (Placebo Comparator): Participants engage in a 20-minute health education session instead of exercise. This arm serves as a non-exercise control to isolate the effects of physical exertion on neuroplasticity. All outcome measures are collected similarly to the exercise groups.
  Interventions: Behavioral: Health education session
- Active Comparator: Moderate-Intensity Aerobic Exercise (Active Comparator): Arm Description: Participants complete a 20-minute cycling session at a moderate workload, surrounding lactate threshold. This condition controls for movement and engagement without advanced metabolic challenge. TMS and motor learning outcomes are assessed pre- and post-intervention.
  Interventions: Behavioral: Moderate Intensity Aerobic Exercise

INTERVENTIONS:
Behavioral: High intensity cycling — Participants cycle on a stationary ergometer at an intensity prescribed to reach their lactate threshold, guided by VO2 max results and lactate sampling. The session lasts approximately 20 minutes and is preceded and followed by TMS assessments and a structured motor learning task. This condition is designed to evaluate the effect of exercise-induced metabolic stress on cortical inhibition and motor learning.
  Other Names: HIIT
  Arms: Aerobic Exercise at Lactate Threshold
Behavioral: Low-intensity cycling — Participants perform 20 minutes of cycling at a light workload below their lactate threshold. Exercise intensity is individualized using heart rate and perceived exertion (Borg RPE scale), avoiding significant metabolic activation. TMS and motor learning are assessed pre- and post-exercise. This condition serves as an active comparator to assess the impact of exercise intensity.
  Other Names: MICT
  Arms: Low-Intensity Aerobic Exercise
Behavioral: Health education session — Participants receive a 20-minute session of health education content (e.g., wellness, healthy aging). No exercise is performed. Participants undergo TMS and motor learning testing before and after the session. This condition is used to control for attention and cognitive engagement without physical activity.
  Other Names: Education
  Arms: Education Control
Behavioral: Moderate Intensity Aerobic Exercise — Participants cycle on a stationary ergometer at an intensity prescribed to surround, but not exceed their lactate threshold, guided by VO2 max results and lactate sampling. The session lasts approximately 20 minutes and is preceded and followed by TMS assessments and a structured motor learning task. This condition is designed to evaluate the effect of moderate exercise-induced metabolic stress on cortical inhibition and motor learning.
  Arms: Active Comparator: Moderate-Intensity Aerobic Exercise

SUMMARY:
The AMPLIFI study (Adaptive Modulation of Plasticity through Lactate and Fitness Interventions) investigates how short-term aerobic exercise influences brain plasticity and learning in older adults and stroke survivors. The study compares three groups: one performing aerobic cycling at an intensity that elevates lactate levels, one performing low-intensity exercise, and one receiving health education without exercise.

All participants will complete motor learning tasks and undergo brain-stimulation testing using transcranial magnetic stimulation (TMS) to assess how well the brain responds to training. The goal is to understand whether different types of exercise can improve brain function, movement, and memory, and how the body's response to exercise (like lactate levels) might support brain health.

This research may help identify low-cost, non-invasive interventions-such as targeted exercise-that improve motor and cognitive outcomes in aging and stroke recovery.

DETAILED DESCRIPTION:
The AMPLIFI study is a mechanistic clinical trial designed to investigate the neurophysiological effects of acute aerobic exercise on cortical plasticity and motor learning in older adults and individuals with chronic stroke. Participants are randomized into one of three groups: (1) moderate-to-high intensity aerobic exercise at lactate threshold, (2) moderate intensity aerobic exercise, (3) low-intensity aerobic exercise, or (4) education-only control.

The primary outcome measure is cortical inhibition, assessed using transcranial magnetic stimulation (TMS) measures including short-interval intracortical inhibition (SICI), long-interval intracortical inhibition (LICI), and intracortical facilitation (ICF). Secondary outcomes include performance on upper extremity motor tasks, measures of verbal and executive function, and blood lactate levels.

Participants complete three sessions over 2-3 weeks, including baseline assessments, VO2 max testing, multiple blood draws, and cognitive and motor testing. The exercise intervention is delivered via stationary cycling at intensities tailored using individual VO2 max data and lactate monitoring. Genetic and biochemical assays will be performed on blood samples to explore associations between metabolic and neural response.

This study will clarify how lactate-related exercise intensity impacts cortical inhibition and whether those effects support improvements in motor learning. Findings may help define the mechanisms by which exercise promotes neuroplasticity and support individualized rehabilitation strategies for aging and post-stroke populations.

ELIGIBILITY:
Inclusion Criteria:

For All Participants:

* Able to provide informed consent
* Right-handed (for TMS consistency)
* English-speaking
* Clearance for moderate-intensity aerobic exercise
* Able to safely sit and pedal a stationary cycle ergometer
* No contraindications to TMS (e.g., no metal in skull, pacemakers, or seizure history)

Younger Adults (18-35):

* No history of neurological or psychiatric conditions
* Not currently on medications that affect the central nervous system

Older Adults (60-85):

* No diagnosis of dementia
* Independent in activities of daily living
* No stroke history

Stroke Survivors (40-85):

* At least 6 months post-stroke (chronic phase)
* Medically stable and cleared for aerobic exercise
* Able to engage in motor learning task (with or without hemiparetic adaptations)

Exclusion Criteria:

* History of epilepsy or seizures
* Current substance abuse or uncontrolled psychiatric disorder
* Severe cardiovascular disease or unstable medical condition
* Pregnancy
* Contraindications to TMS or exercise testing (e.g., implanted neurostimulators, severe hypertension)
* Participation in another interventional trial within the past 30 days

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-04-14 (Estimated); Primary Completion 2029-09-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Motor Learning Performance (12-Digit Serial Reaction Time Task) | Baseline, Day 2, Day 3, Day 4, and Day 5
  Motor learning is assessed using the 12-digit Serial Reaction Time Task (SRTT), a computer-based measure of implicit motor sequence learning. Participants respond to visual cues by pressing buttons in a fixed or random sequence. Learning is quantified by changes in reaction time and accuracy across structured and unstructured trials. A learning index is derived by comparing performance between patterned (learning) and random sequences.

SECONDARY OUTCOMES:
Change in Long-Interval Intracortical Inhibition (LICI) | Baseline, Day 5
  LICI is measured using a 100 ms interstimulus interval to assess GABA<sub>B</sub>-mediated inhibition. Recorded before and after each intervention session.
Change in Intracortical Facilitation (ICF) | Baseline, Day 5
  ICF is assessed using paired-pulse TMS with a 10-15 ms interstimulus interval to evaluate cortical excitability.
Change in Blood Lactate Concentration | Day 2, Day 3, Day 4
  Measured via fingerstick blood samples pre-, mid-, and post-exercise.
Change in Executive Function (D-KEFS Verbal Fluency and Stroop Tests) | Day 1 and Day 5
  Executive function neuropsychological tests.

CONTACTS AND LOCATIONS:
Overall Officials: Keith McGregor, PhD, Principal Investigator — Keith McGregor
Locations (1):
- CH19 933 19th St S, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
No, not beyond the original research team.